CLINICAL TRIAL: NCT03261804
Title: Relation Between Internal Vaginal Douching and Vaginal Infections in Intrauterine Contraceptive Device Users
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Alaaeldin Mahmoud Youssef, Lecturer of Obstetrics and Gynaecology, Women Health Hospitals, Assiut University, Assiut University
Other Study IDs: VD in IUD users
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Vaginal Infection
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I:internal vaginal douching users
  Interventions: Behavioral: relation between vaginal douching and vaginal infection
- Group II: none internal vaginal douching users
  Interventions: Behavioral: relation between vaginal douching and vaginal infection

INTERVENTIONS:
Behavioral: relation between vaginal douching and vaginal infection — personal hygiene including performing external or Internal vaginal douching, how she is performing this douching (by hand, water, jet, pump), how frequent and why they perform this internal vaginal douche.

SUMMARY:
To determine the effect of performing internal vaginal douching on the frequency and severity and type of vaginal infections in IUD users

DETAILED DESCRIPTION:
The actual frequency of infectious vaginitis is difficult to determine, due to numerous confounding factors, such as a high asymptomatic rate, inaccurate self-diagnosis and treatment, and population dependence. In the USA, the prevalence of cervicovaginal infections was 29.1% and that bacterial vaginosis was frequently found 19.7% among IUDs users 6 months after insertion.

Vaginal douching (VD) is the process of intravaginal cleansing with any type of liquid solution. Douching is a common practice among women all over the world and is used for personal hygiene. Studies in the USA showed that about 37% of US women in reproductive age (15-44 Y) reported regular VD. The performance of this habit varied between different ethnic groups and different socioeconomic levels. In a Turkish study, VD reported to be performed by 91.6% of women living in rural areas.

There are cultural believes that VD is necessary for good hygiene. Other motives for douching are to clean the vagina after the end of menses or before and/or after sexual intercourse, to prevent or ameliorate an odor, to prevent or treat vaginal symptoms such as itching and discharge. Other factors contribute to a woman's decision to douche her vagina like the influence of patients' mothers, friends, and relatives. Some others consider VD as religious duty to be able to pray after menses or sexual intercourse.

Previous studies have pointed to reproductive health hazards of VD. Women who perform this habit were 1.2 to 5.1 times more likely to develop bacterial vaginosis (BV); 1.6 -1.9 times more likely to experience a preterm labor (PTL). Women who adopt this habit were twice likely to develop cancer cervix; 1.7 times more likely to have sexually transmitted infections (STIs). Moreover, VD performers have 73% increased risk of pelvic inflammatory disease (PID) and are 1.5 times more likely to develop endometritis.

The intrauterine device (IUD) is the most widely used method of contraception because of its safety and cost-effective benefit. Over 100 million women are now using this device. However, the number of user is still much less than expected. This probably due to the doubt about complications from IUD, the most common medical reasons for early discontinuation of IUD are bleeding and/or pain along with genital infections.

Many women who have vaginitis generally complain of some combination of discharge, odor, irritation, and itch. The most common causes of vaginitis in premenopausal group were bacterial vaginosis, vaginal candidiasis and trichomoniasis. Previous studies showed that copper IUD caused a change in the cervicovaginal flora that resulted in the predominance of anaerobic species. These alterations may affect vaginal health and cause more vaginal infection and symptoms for example itching, soreness and abnormal discharge.

ELIGIBILITY:
Inclusion Criteria:

* 1- Women currently using cu IUD for at least 6 months before the study 2-Within the age 18-48 years 3-Accept to participate in the study

Exclusion Criteria:

* 1-Woman who are using a contraceptive method other than IUD 2-Any other endocrinal disease like DM , thyroid ……etc 3- Patient under chemotherapy for treatment of cancer 4- antibiotic and Steroid users 5-inperfect IUD place

Ages: 18 Years to 48 Years | Sex: Female
Age Groups: Adult
Study Population: Family planning and population growth problems
Sampling Method: Non-Probability Sample
Enrollment: 604 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
frequency of vaginal infections in IUD user | 18 months
  Compare frequency of vaginal infections in IUD user who perform internal vaginal douching with not perform internal vaginal douching

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A YOUSSEF, M.D, Principal Investigator — Assiut University
Locations (1):
- Women's Health Hospital, Assiut University, Asyut, Egypt

REFERENCES:
- [Result] Ferraz do Lago R, Simoes JA, Bahamondes L, Camargo RP, Perrotti M, Monteiro I. Follow-up of users of intrauterine device with and without bacterial vaginosis and other cervicovaginal infections. Contraception. 2003 Aug;68(2):105-9. doi: 10.1016/s0010-7824(03)00109-4. PMID 12954522
- [Result] Martino JL, Vermund SH. Vaginal douching: evidence for risks or benefits to women's health. Epidemiol Rev. 2002;24(2):109-24. doi: 10.1093/epirev/mxf004. No abstract available. PMID 12762087
- [Result] Zhang J, Thomas AG, Leybovich E. Vaginal douching and adverse health effects: a meta-analysis. Am J Public Health. 1997 Jul;87(7):1207-11. doi: 10.2105/ajph.87.7.1207. PMID 9240115
- [Result] Zhang J, Hatch M, Zhang D, Shulman J, Harville E, Thomas AG. Frequency of douching and risk of bacterial vaginosis in African-American women. Obstet Gynecol. 2004 Oct;104(4):756-60. doi: 10.1097/01.AOG.0000139947.90826.98. PMID 15458898
- [Result] Hutchinson KB, Kip KE, Ness RB; Gynecologic Infection Follow-Through (GIFT) Investigators. Vaginal douching and development of bacterial vaginosis among women with normal and abnormal vaginal microflora. Sex Transm Dis. 2007 Sep;34(9):671-5. doi: 10.1097/01.olq.0000258435.34879.da. PMID 17413534
- [Result] Luong ML, Libman M, Dahhou M, Chen MF, Kahn SR, Goulet L, Seguin L, Lydon J, McNamara H, Platt RW, Kramer MS. Vaginal douching, bacterial vaginosis, and spontaneous preterm birth. J Obstet Gynaecol Can. 2010 Apr;32(4):313-320. doi: 10.1016/S1701-2163(16)34474-7. PMID 20500937
- [Result] Fonck K, Kaul R, Keli F, Bwayo JJ, Ngugi EN, Moses S, Temmerman M. Sexually transmitted infections and vaginal douching in a population of female sex workers in Nairobi, Kenya. Sex Transm Infect. 2001 Aug;77(4):271-5. doi: 10.1136/sti.77.4.271. PMID 11463927
- [Result] Rew L. Vaginal douching increased risk of sexually transmitted infections in high-risk adolescents. Evid Based Nurs. 2009 Jul;12(3):88. doi: 10.1136/ebn.12.3.88. No abstract available. PMID 19553425
- [Result] Kanat-Pektas M, Ozat M, Gungor T. The effects of TCu-380A on cervicovaginal flora. Arch Gynecol Obstet. 2008 May;277(5):429-32. doi: 10.1007/s00404-007-0496-0. Epub 2007 Oct 31. PMID 17972087
- [Result] Haukkamaa M, Stranden P, Jousimies-Somer H, Siitonen A. Bacterial flora of the cervix in women using an intrauterine device. Contraception. 1987 Nov;36(5):527-34. doi: 10.1016/0010-7824(87)90004-7. PMID 3447813